CLINICAL TRIAL: NCT01789554
Title: The Response to Urgent Mobile Message for Bystander Activation (RUMBA) Trial - The Use of Mobile Phone Positioning for Dispatch of Bystanders to Out of Hospital Cardiac Arrest.
Brief Title: The Use of Mobile Phones in Out of Hospital Cardiac Arrest to Increase Bystander CPR
Acronym: RUMBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Leif Svensson, Professor, Karolinska Institutet
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: RUMBA2013
Record Dates: First submitted 2013-02-06; First posted 2013-02-12 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Out-of-Hospital Cardiac Arrest; Death, Sudden, Cardiac; Heart Diseases; Ventricular Fibrillation
Keywords: Out of hospital cardiac arrest; Cardiopulmonary resuscitation; Bystander CPR; Mobile phone positioning system
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Death, Sudden, Cardiac; Heart Diseases; Ventricular Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MLS dispatch for bystander CPR (Experimental): When an alarm call of a suspected OHCA suspected is received by the EMS dispatch operator a Mobile positioning system (MPS) is activated. The MPS uses the mobile phone network to geographically locate all lay volunteers connected to a tailored mobile phone service called mobile life saver (MLS). The MPS then locates all lay volunteers within a pre defined radius from the suspected OHACA an alerts them with a computer generated voice call and an sms containing data about were about were the suspected OHCA is located. A map is also sent in order to make route finding easy.
  Interventions: Other: MLS dispatch for bystander CPR
- NO MLS dispatch for bystander CPR (No Intervention): No activation of mobile positioning system to locate and recruit lay responders to nearby OHCAs

INTERVENTIONS:
Other: MLS dispatch for bystander CPR
  Arms: MLS dispatch for bystander CPR

SUMMARY:
Death from cardiac disease is one of the most common causes of death in the western world. The majority of these deaths takes place outside hospital as sudden cardiac death. However, with immediate (within minutes) actions such as cardiopulmonary resuscitation (CPR) and defibrillation many lives would be saved. CPR is a key factor to increase survival from Out of Hospital Cardiac Arrest (OHCA). CPR buys time by supporting the brain with some circulation in waiting for a defibrillator that can restart the heart. In Sweden about 2,5 million people are trained in CPR. However, only about half of all OHCA victims will get CPR in waiting for ambulance arrival.

The aims of the Response to Urgent Mobile message for Bystander Activation (RUMBA) trial is to try a new way of logistics to increase bystander CPR by recruiting lay volunteers to nearby OHCAs via their mobile phones.

Hypothesis: By dispatching lay volunteers to nearby OHCAs with mobile phone technology bystander CPR may increase from 50% to 62,5 %

DETAILED DESCRIPTION:
Survival from out-of-hospital cardiac arrest (OHCA) is generally low, about 5-10%, with the exception of a few controlled settings (casinos, airports and some cities). The poor prognosis of OHCA is mainly explained by long time intervals between cardiac arrest, cardiopulmonary resuscitation (CPR) and defibrillation. To increase bystander actions and to decrease time to defibrillation substantial resources have been put into CPR educational campaigns and in recent years into the spread of automated external defibrillators (AEDs) in public venues. Still, the vast majority of the public with CPR training will never use their skills in real life. Mobile phone technology offers the possibility to locate single mobile phone users at any given moment. If designated lay responders immediately can be identified and recruited to the scene of nearby suspected OHCAs bystander CPR, CPR quality and finally survival might be increased.

Mobile phone positioning and dispatching of lay responders:

Tailored mobile phone services that use MPS to locate selected mobile phone users can be developed for different purposes. A computer-based application for mobile phone positioning and dispatch of lay responders is developed for the purpose of this study and is referred to as the Mobile Lifesaver Service (MLS). All participants connected to the MLS are called Mobile Responders (MRs). The MLS acts as an interface between the emergency medical service (EMS) data system and the MPS. The MLS handles the localisation and dispatching of MRs based on the data present in the EMS data system. The location of all incoming calls to all dispatch centres in Sweden is determined automatically.

When the dispatcher receives an emergency call from a witness of a suspected OHCA the dispatcher activates the MLS in parallel with standard EMS. When the MLS is activated it uses the MPS to compare the current geographical position of all MRs connected to the MLS with the position of the incoming emergency call of the suspected cardiac arrest. If one or more MRs is present within a radius of 500 m (optional) from the suspected arrest the MRs receives a cardiac arrest alert with a computer generated phone call and a text message (i.e. SMS = short message system) with information about the place of the suspected cardiac arrest. A map for finding the way to the suspected OHCA is also sent. Additional information can, if needed, be sent to the MRs.

For further details see "Mobile phone technology identifies and recruits trained citizens to perform CPR on out-of-hospital cardiac arrest victims prior to ambulance arrival." Ringh M, Fredman D, Nordberg P, Stark T, Hollenberg J. Resuscitation. 2011 Dec;82(12):1514-8.

Data from earlier non randomized pilot studies in urban Stockholm has shown that CPR was performed by MLS dispatched lifesavers prior to ambulance, firefighters and police in about 20 % of all cases of true OHCAs.

The hypothesis is that bystander CPR in Stockholm County can be increased from 50 % to 62,5% if the MLS is used. An estimated number of 6000 MR needed is based on earlier pilot studies.

The current proportion of bystander CPR is derived from OHCA registry data but is uncertain.

A safety and efficacy analyze will be made at approximately 200 true OHCA cases.

A ethical and safety board and log for adverse events will be set up.

ELIGIBILITY:
Inclusion Criteria:

* All suspected OHCAs in Stockholm County
* All EMS treated out of hospital cardiac arrest in Stockholm County were the mobile positioning system is triggered

Exclusion Criteria:

* Traumatic OHCA
* Children under 8 years of age
* Suicide
* Intoxications
* Obvious signs of death
* Do not resuscitate orders (DNR)

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Bystander CPR by trained bystander before arrival of ambulance, firefighters or police | Within 1 hour from randomization
  Bystander CPR is defined as CPR by trained laymen in Out of hospital Cardiac Arrest patients before arrival of ambulance, firefighters or police and this only in OHCA patients were care is continued by ambulance crew. CPR in cases showing obvious signs of death are excluded. Telephone assisted CPR by untrained laymen is not accounted for as bystander CPR.

SECONDARY OUTCOMES:
OHCAs were lay volunteers dispatched by the mobile positioning system arriving prior to ambulance | Within 1 hour from randomization
  The proportion of mobile phone dispatched lay volunteers arriving prior to ambulance at the scene of the OHCA
Time of bystander CPR before arrival of ambulance, firefighters or police | Within 1 hour from randomization
  The time of bystander CPR performed by mobile phone dispatched lay volunteer before arrival of ambulance, firefighters or police
Rhythm on first ECG | Within 1 hour from randomization
  Defined as the cardiac rhythm recorded on first ECG. Either Ventricular fibrillation/pulseless ventricular tachycardia (VF/VT) or asystole/pulseless electrical activity If defibrillation = VF/VT
Return of spontaneous circulation (ROSC) | Within 3 hours from randomization
  The return of circulation after successful CPR that can be felt by palpable puls or blod pressure that can be measured
Admitted alive | 24 hours after hospital admission
  Admitted from Emergency to hospital ward (usually ICU) and alive 24 h after admission
Alive after 1 month Cerebral Performance Categories (CPC) 1-2 | From OHCA and 30 days
  Alive after 30 days with CPC score 1-2.
  Description:
  The Cerebral Performance Categories (CPC) are used to describe neurological outcome. A CPC of 1 or 2 is considered "neurologically intact."
  * Good cerebral performance: little to no deficit.
  * Moderate cerebral disability: capable of independent activities of daily life
  * Severe cerebral disability: conscious, but dependent on others for daily support
  * Coma or vegetative state
  * Death or brain death
Alive after 1 month CPC 1-2 | From OHCA and 90 days
  Alive after 90 days with CPC score 1-2.

CONTACTS AND LOCATIONS:
Overall Officials: Leif Svensson, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Department of Cardiology Södersjukhuset, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Derived] Ringh M, Rosenqvist M, Hollenberg J, Jonsson M, Fredman D, Nordberg P, Jarnbert-Pettersson H, Hasselqvist-Ax I, Riva G, Svensson L. Mobile-phone dispatch of laypersons for CPR in out-of-hospital cardiac arrest. N Engl J Med. 2015 Jun 11;372(24):2316-25. doi: 10.1056/NEJMoa1406038. PMID 26061836